CLINICAL TRIAL: NCT07073885
Title: The Effect of Ultra-Low Tidal Volume Ventilation on Mechanical Power in Coronary Artery Bypass Graft Surgery
Brief Title: Effect of Ultra-Low Tidal Volume on Mechanical Power During Heart Bypass Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Esma Karaarslan, Medical Doctor (MD), Department of Anesthesiology and Reanimation, Konya City Hospital, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CABGO-MP
Record Dates: First submitted 2025-07-02; First posted 2025-07-18 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ULTV (Experimental): Participants in this group will continue to receive mechanical ventilation after aortic cross-clamping during cardiopulmonary bypass (CPB). Ventilation will be provided in volume-controlled mode with a tidal volume of 3-4 mL/kg ideal body weight, respiratory rate of 12-14 breaths/min, 5 cm H₂O PEEP (Positive End-Expiratory Pressure), and 50% FiO₂.
  .
  Interventions: Other: Ultra-Low Tidal Volume Ventilation
- Apnea Group (Active Comparator): After the application of the aortic cross-clamp, mechanical ventilation will be discontinued, and apnea will be maintained.
  Interventions: Other: Apnea Group

INTERVENTIONS:
Other: Ultra-Low Tidal Volume Ventilation — Ventilation continued during CPB using volume-controlled mode with ultra-low tidal volume (3-4 mL/kg IBW(Ideal Body Weight)), 12-14 breaths/min, 5 cm H₂O PEEP, and 50% FiO₂.
  Arms: Group ULTV
Other: Apnea Group — In this group, mechanical ventilation will be discontinued after aortic cross-clamping during CPB, and apnea will be maintained throughout the bypass period.
  Arms: Apnea Group

SUMMARY:
The goal of this clinical trial is to evaluate whether ultra-low tidal volume (ULTV) ventilation during cardiopulmonary bypass (CPB) can reduce mechanical power (MP) and improve postoperative respiratory outcomes in adult patients undergoing elective coronary artery bypass graft (CABG) surgery.

The main questions it aims to answer are:

Does ULTV ventilation during CPB result in lower intraoperative mechanical power compared to apnea?

Can ULTV ventilation reduce extubation time and ICU (Intensive Care Unit) stay and improve the PaO₂/FiO₂ ratio (Partial Pressure of Arterial Oxygen / Fraction of Inspired Oxygen Ratio)?

Researchers will compare patients receiving ULTV ventilation to those undergoing apnea after aortic cross-clamping to assess the effects on mechanical power and postoperative outcomes.

Participants will:

Be randomized to either ULTV ventilation or apnea group

Undergo standard general anesthesia and CABG surgery

Have mechanical power measured at three time points (pre-CPB, post-CPB, and ICU pre-extubation)

Have arterial blood gases evaluated for PaO₂/FiO₂ ratios

Be monitored for extubation time and ICU length of stay

This study aims to generate evidence that could inform safer and more protective intraoperative ventilation strategies during cardiac surgery.

DETAILED DESCRIPTION:
This is a prospective, randomized, assessor-blinded, single-center clinical trial designed to evaluate the effects of ultra-low tidal volume (ULTV) ventilation on intraoperative mechanical power (MP) and postoperative pulmonary outcomes in patients undergoing elective coronary artery bypass graft (CABG) surgery with cardiopulmonary bypass (CPB).

After obtaining informed consent, eligible adult patients (ASA II-IV) scheduled for elective CABG will be randomly assigned to one of two groups:

ULTV Group: Ventilation will be continued after aortic cross-clamping using volume-controlled ventilation with a tidal volume of 3-4 mL/kg ideal body weight, 12-14 breaths per minute, 5 cm H₂O PEEP, and 50% FiO₂.

Apnea Group: Mechanical ventilation will be discontinued after aortic cross-clamping, and patients will remain apneic during CPB.

Mechanical power will be calculated using a validated surrogate formula and measured at three key time points: pre-CPB (baseline), post-CPB (before ICU transfer), and at the 3rd postoperative hour in the ICU (before extubation). Arterial blood gases will be obtained to determine PaO₂/FiO₂ ratios at these time points and 24 hours post-extubation.

Secondary outcomes include extubation time and length of ICU stay.

This study aims to generate evidence supporting the potential protective effects of continued low-volume ventilation during CPB, with a focus on reducing ventilator-induced lung injury by limiting mechanical power and preserving alveolar integrity.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex aged over 18 years
* Patients classified as ASA II-IV
* Patients scheduled for elective CABG

Exclusion Criteria:

* Presence of severe COPD
* Uncontrolled bronchial asthma
* Decompensated heart failure (NYHA class III-IV)
* Pulmonary hypertension
* History of lung surgery
* Morbid obesity (BMI >35)
* Emergency surgery cases
* Patients who decline to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Mechanical Power | MP Measurements (Mechanical Power) MP 1: Baseline (after intubation and before surgical incision) MP 2: At the end of surgery (prior to ICU admission) MP 3: Postoperative 3rd hour in ICU (prior to extubation)
  Primary Aim Measurements Calculation of Mechanical Power (MP)
  Several methods exist for measuring MP. In this study, a simplified and validated method will be employed. The formula is expressed as follows:
  MP (J/min) = 0.098 × RR × Vt × (PEEP + ½[Pplat - PEEP] + [Ppeak - Pplat]) (RR: Respiratory Rate, Vt : Tidal Volume, PEEP: Positive End-Expiratory Pressure, Pplat: Plateau Pressure, Ppeak: Peak Inspiratory Pressure).
  Thus, MP is calculated as the product of the work per individual breath (volume × pressure) multiplied by the respiratory rate. Primary evaluation parameters will be computed using ventilator settings, with three consecutive measurements taken and averaged for accuracy.

SECONDARY OUTCOMES:
extubation time | From the end of surgery until the time of tracheal extubation, assessed up to 24 hours postoperatively.
  Extubation time is defined as the duration (in hours) from the end of surgery to the time of tracheal extubation.
duration of intensive care unit (ICU) stay. | From ICU admission following surgery until ICU discharge, assessed up to 7 days postoperatively.
  Defined as the number of calendar days the patient remains in the intensive care unit (ICU) following surgery, until transfer to the general ward. Data will be collected daily during ICU stay.
PaO₂/FiO₂ ratio. | 1. Baseline (after intubation, before surgical incision) 2. At the end of surgery (prior to ICU admission) 3. Postoperative 3rd hour in ICU (prior to extubation) 4. 24 hours after extubation
  PaO₂/FiO₂ ratios will be calculated from arterial blood gas samples obtained at four predefined time points: after intubation and before surgical incision (preoperative baseline), at the end of surgery (prior to ICU admission), at the 3rd postoperative hour in the ICU (before extubation), and at the 24th hour following extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Esma karaarslan, MD, Principal Investigator — Konya City Hospital
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
maybe, we can share all info after finish the study
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The exact time frame for data sharing will be determined after the study is completed and the results are published.
Access Criteria: we can share the data by using e-mail